CLINICAL TRIAL: NCT02532088
Title: Modulating Effects of Oil Palm Phenolics in Subjects With Pre-diabetes
Acronym: PREDOPP
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Project terminated
Sponsor: Universiti Sains Malaysia (Other)
Collaborators: Malaysia Palm Oil Board (Other Government); Clinical Research Centre, Malaysia (Other)
Responsible Party: Principal Investigator, Yuen Kah Hay, Professor, Dr., Universiti Sains Malaysia
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PREDOPP-21100
Record Dates: First submitted 2015-08-10; First posted 2015-08-25 (Estimated); Last update posted 2021-10-06 (Actual); Status verified 2021-09

CONDITIONS: Prediabetes
MeSH Terms: conditions — Prediabetic State

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Oil Palm Phenolics (Active Comparator): 500 mg gallic acid equivalent (GAE), twice daily, 12 months
  Interventions: Dietary Supplement: Oil Palm Phenolics
- Placebo (Placebo Comparator): Placebo
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Oil Palm Phenolics — Palm fruit derived phenolics compound
  Arms: Oil Palm Phenolics
Dietary Supplement: Placebo — Placebo
  Arms: Placebo

SUMMARY:
Study reported that providing Oil Palm Phenolics to Nile rats blocked diabetes progression in this spontaneous diabetes model. The present study aims to determine the beneficial effects of Oil Palm Phenolics in subjects with pre-diabetes.

DETAILED DESCRIPTION:
Recent studies suggest the potential of polyphenols as a supplementary treatment to delay or prevent the onset of diabetes owing to their biological properties. Polyphenols are natural phytochemical compounds found in fruits and vegetables. The most common group of phenolic compounds in our diet are phenolic acids and flavonoids. The two main classes are hydroxybenzoic acid derivatives and hydroxycinnamic acid derivatives. The anti-hyperglycemic property of polyphenols is mainly contributed by the reduction of dietary carbohydrate absorption through intestines, improvement of β-cell function and insulin action, stimulation of insulin secretion, modulation of the enzymes involved in glucose metabolism, anti-oxidative and anti-inflammatory effects.

The key enzymes responsible for the digestion of dietary carbohydrates to glucose are α-glucosidase and α-amylase. One of the most well-known properties of polyphenols especially phenolic acids on carbohydrate metabolism is the inhibition of these enzymes. Some investigations have shown that polyphenols are also able to regulate postprandial glycemia and inhibit the development of glucose intolerance by a facilitated insulin response and increased secretion of glucose-dependent insulinotropic polypeptide (GIP) and glucagonlike polypeptide-1 (GLP-1). In addition, polyphenols are able to regulate the key pathways involved in carbohydrate metabolism and hepatic glucose homeostasis. These include glycolysis, glycogenesis and gluconeogenesis, which are usually impaired in diabetes.

The current study focuses on the glucose-controlling properties of phenolic compounds extracted from oil palm (Elaeis guineensis), a high oil-producing tropical plant that also rich in phytochemicals. The major phenolic components in OPP are identified as caffeoylshikimic acid, protocatechuic acid and p-hydroxybenzoic acid. OPP has been found to exert various positive health effects parallel to the well-established physiological benefits of polyphenols. It has been shown that OPP protects against early type 2 diabetes and encouraging results suggest its role in modulating the development of diabetes. The current study aims to investigate and determine the effects of oil palm phenolics (OPP) on the blood glucose control in pre-diabetics.

ELIGIBILITY:
Inclusion Criteria:

* Subject with "pre-diabetes", i.e. fasting plasma glucose level of more than 5.6 mmol/L and less than 7.0 mmol/L; or 2-hr plasma glucose load level of more than 7.8 mmol/L and less than 11.0 mmol/L.
* Subjects or his/her legally acceptable representative is willing to provide written informed consent.

Exclusion Criteria:

* Subject with terminal cancer.
* Subject with renal failure (serum creatinine more than 200 umol/L).
* Subject with significant liver impairment (liver function test of 5 times more than the upper limit level).
* Subject with severe dementia and psychosis.
* Subject requires of long term corticosteroid treatment for the underlying disease such as connective tissue disorder.
* Subject with hemoglobinopathy or anemia.
* Subject underwent splenectomy or suffered from splenomegaly.
* Subject with pre-existing cardiovascular disease.
* Subject with chronic substance abuse such as chronic alcoholism or chronic opiate usage.
* Female subject of childbearing potential unless subject underwent bilateral tubal ligation, bilateral oophorectomy or hysterectomy previously.
* Subject with other significant uncontrolled medical illnesses that may interfere with drug administration or interpretation of results.
* Subject who have been included in any other clinical trial within the previous 3 months.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-05 (Estimated); Primary Completion 2021-06 (Estimated); Study Completion 2021-09 (Estimated)

PRIMARY OUTCOMES:
Blood Glucose Level | 12 months
  1. Serum Glycosylated Haemogoblin (<5.7% indicates healthy, 5.7% - 6.4% indicates prediabetes, >6.5% indicates diabetes)
  2. Plasma glucose level of oral glucose tolerance test (<7.8 mmol/L indicates healthy, 7.8 mmol/L - 11 mmol/L indicates prediabetes, >11 mmol/L indicates diabetes)
  3. Fasting plasma glucose level (<5.6 mmol/L indicates healthy, 5.6 mmol/L - 6.9 mmol/L indicates prediabetes, >6.9 mmol/L indicates diabetes)

SECONDARY OUTCOMES:
Insulin Sensitivity | 12 months
  Model-derived Oral Glucose Insulin Sensitivity (OGIS) Index will be calculated using weight (kg), height (cm), glucose (mmol/L) and insulin (pmol/L).
Lipid profile | 12 months
  Total cholesterol, Low-density lipoprotein, High-density lipoprotein, Triglycerides
Global Assessment of Efficacy | 12 months
  Very good, good, no change, unsatisfactory and very unsatisfactory
Beta Cell Function | 12 months
  Homeostatic Model Assessment (HOMA2-B) to determine beta cell function

CONTACTS AND LOCATIONS:
Overall Officials: Kah Hay Yuen, PhD, Principal Investigator — Universiti Sains Malaysia
Locations (1):
- Seberang Jaya Hospital, Seberang Jaya, Pulau Pinang, Malaysia

IPD SHARING:
Plan to Share IPD: No